CLINICAL TRIAL: NCT00024011
Title: A Phase II Study of PS-341 in the Treatment of Metastatic Malignant Melanoma
Brief Title: PS-341 in Treating Patients With Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02409; MC007A; N01CM17104 (NIH); CDR0000068883 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-09-13; First posted 2004-02-06 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Bortezomib

ARMS (1):
- Treatment (bortezomib) (Experimental): Patients receive PS-341 IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of PS-341 in treating patients who have metastatic malignant melanoma. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the progression-free survival at 18 weeks and overall survival of patients with metastatic malignant melanoma treated with PS-341.

II. Determine the objective response rate of patients treated with this drug. III. Correlate p27 levels in tumor tissue with objective response rate in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive PS-341 IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3-6 months for up to 2 years after registration.

PROJECTED ACCRUAL: A total of 22-50 patients will be accrued for this study within 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic malignant melanoma
* Measurable disease defined as at least one lesion whose longest diameter can be accurately measured as >= 2.0 cm
* Absolute neutrophil count (ANC) >= 1500/uL
* PLT >= 100,000/uL
* Total bilirubin =< 2.5 x institutional upper normal limit (UNL)
* AST =< 2.5 x UNL
* Creatinine =< 1.5 x UNL or calculated creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels > 1.5 x UNL using the Cockcroft-Gault formula
* Life expectancy of >= 3 months
* ECOG performance status 0 or 1
* Capable of understanding the investigational nature, potential risks and benefits of the study and willing to sign the written informed consent document

Exclusion Criteria:

* Any of the following:

  * Any prior chemotherapy
  * Immunotherapy =< 4 weeks prior to study entry
  * Biologic therapy =< 4 weeks prior to study entry
  * Radiation therapy =< 4 weeks prior to study entry
  * Failure to fully recover from adverse effects of prior therapies regardless of interval since last treatment
  * Other concurrent chemotherapy, immunotherapy, radiotherapy, or any other therapy or supportive care considered investigational
* Known brain metastases requiring active treatment; NOTE: these patients are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PS-341
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris, cardiac arrhythmia
  * Psychiatric illness that would limit compliance with study requirements
* HIV-positive patients receiving combination anti-retroviral therapy; NOTE: patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; these patients are excluded from the study because of possible pharmacokinetic interactions with PS-341; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, subcutaneous implants, intrauterine device [IUD], abstinence, etc.)
  * NOTE: this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown
* Only non-measurable disease, including lesions not clearly measurable in one dimension, small lesions (longest diameter < 20 mm), and truly non-measurable lesions, which include the following as per RECIST criteria:

  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Inflammatory breast disease
  * Lymphangitis cutis/pulmonis
  * Abdominal masses that are not confirmed and followed by imaging techniques
  * Cystic lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-07; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are progression-free | 18 weeks
  Confidence intervals for the true success proportion will be calculated.

SECONDARY OUTCOMES:
Objective response is defined by the Response Evaluation Criteria in Solid Tumors (RECIST) in terms of tumor/lesion size and change | Up to 2 years
Overall survival | Time from registration to death due to any cause, assessed up to 2 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States